CLINICAL TRIAL: NCT06255392
Title: Randomized, Open, Controlled, Multicenter Phase III Clinical Study of Fluzoparib in Combination With Apatinib Versus Investigator-Selected Chemotherapy for HRD-Positive/HER2-negative Advanced Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-1016-04
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Fludzoparib" and Anti-angiogenic; HRD-positive/HER2-negative Advanced Breast Cancer
MeSH Terms: interventions — fluzoparib; apatinib; Capecitabine; Vinorelbine; eribulin; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluzoparib Combined With Apatinib (Experimental): Fluzoparib combined with Apatinib group: Fluzoparib capsules oral +Apatinib Mesylate oral; each treatment cycle defined as 3 weeks (21 days).
  Interventions: Drug: Fluzoparib; Drug: Apatinib Mesylate
- Chemotherapy selected by the investigator (Active Comparator): Control group: Control group: patients receive oral Capecitabine tablets, Vinorelbine Tartrate Capsules, or use intravenous Paclitaxel for Injection (Albumin Bound), Gemcitabine Hydrochloride for Injection, or other drugs selected by the investigator.
  Interventions: Drug: Capecitabine tablets; Drug: Vinorelbine Tartrate Oral; Drug: Eribulin mesylate injection; Drug: Gemcitabine Hydrochloride; Drug: Paclitaxel-albumin

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib capsules appropriate dose oral, each treatment cycle defined as 3 weeks (21 days).
  Arms: Fluzoparib Combined With Apatinib
Drug: Apatinib Mesylate — Apatinib Mesylate oral; each treatment cycle defined as 3 weeks (21 days).
  Arms: Fluzoparib Combined With Apatinib
Drug: Capecitabine tablets — Capecitabine tablets, reasonable dosage with reference to guidelines, each treatment cycle defined as 3 weeks (21 days).
  Arms: Chemotherapy selected by the investigator
Drug: Vinorelbine Tartrate Oral — For the first three courses: reasonable dosage with reference to guidelines. After 3 courses of medication, it is recommended to increase the dose of vinorelbine tartrate once a week. Each treatment cycle defined as 3 weeks (21 days).
  Arms: Chemotherapy selected by the investigator
Drug: Eribulin mesylate injection — Eribulin, reasonable dosage with reference to guidelines, each treatment cycle defined as 3 weeks (21 days).
  Arms: Chemotherapy selected by the investigator
Drug: Gemcitabine Hydrochloride — Gemcitabine, reasonable dosage with reference to guidelines, each treatment cycle defined as 3 weeks (21 days).
  Arms: Chemotherapy selected by the investigator
Drug: Paclitaxel-albumin — Paclitaxel-albumin, reasonable dosage with reference to guidelines, each treatment cycle defined as 3 weeks (21 days).
  Arms: Chemotherapy selected by the investigator

SUMMARY:
This study develops a new therapeutic approach for HER2-negative advanced breast cancer patients without precise treatment targets. The trial aims at extending the combination target therapy involving PARP inhibitors and anti-angiogenesis from only BRCA mutation carriers to all patients with homologous recombination repair defects (HRD-positive). The phase III randomized clinical study will investigate the effectiveness of the combination therapy of PARP inhibitor "fludzoparib" and anti-angiogenic "apatinib" in treating HRD-positive/HER2-negative advanced breast cancers.

DETAILED DESCRIPTION:
Breast cancer is the most prevalent malignant tumor in the world, and 30% of breast cancer patients will enter the advanced stage due to treatment failure. 80% of these patients have HER2-negative subtype breast cancer, which has not yet been found the similar target as HER2, with the median survival time of only 6-20 months. In the past, ovarian cancer patients faced the dilemma of poor survival due to the lack of precise targeted therapy. However, through a series of clinical studies, experts in the field of ovarian cancer have successfully expanded the indications of PARP inhibitor-based combination targeted therapy from the small population of BRCA mutation(20%) to the large population of HRD-positive (Homologous recombination deficiency) (50%), which has significantly prolonged the survival time of patients. Because causes other than BRCA mutations can also cause tumor cells to be "HRD" and thus sensitive to PARP inhibitors, so that HRD-positive patients are likely to benefit. The HRD-positive profile of nearly 50% of the patients could be a potential beneficiary of PARP inhibitor-based targeted therapy. The synergistic effect of PARP inhibitor and anti-angiogenic combination therapy has already been confirmed in preliminary cellular experiments and clinical studies related to ovarian cancer. Further cell-based experiments and preclinical studies have also confirmed the feasibility of the combination targeted therapy in the HRD-positive/HER2-negative subtype of breast cancer. Therefore, we intend to further validate the efficacy and safety of the PARP inhibitor fluazoparib in combination with the antiangiogenic abatinib in a Phase III, randomized, controlled clinical study, in order to provide HRD-positive/HER2-negative breast cancer patients with a better choice of precision targeted therapy.

ELIGIBILITY:
Inclusion criteria

The subjects must meet all of the following conditions:

Adult female patients (aged 18 to 70 years) with metastatic breast cancer diagnosed by pathology or imaging; 2) Pathological confirmation of HER2 negative (definition: immunohistochemical result is 0 or + or ++ and in situ hybridization result is negative); 3) The patient's HRD test was positive (definition: BRCA1/2 mutation, or HRD score greater than or equal to 42 points); 4) HR+/HER2- patients who have received endocrine therapy during the metastasis stage; 5) Having received no more than two lines of chemotherapy (or ADC) regimens for metastatic breast cancer in the past; 6) Evaluation of anti-tumor treatment (including chemotherapy /HER2-ADC/TROP2-ADC) for 6-8 cycles to achieve clinical benefit (CR or PR) or SD for 24 weeks or more; 7) ECOG physical condition score ≤2 points, and the expected survival period is no less than 3 months; 8) At least one measurable lesion was found in the imaging examination within 2 weeks before enrollment. Or simple bone metastasis lesion; 9) At the time of enrollment, the previous treatment-related toxicity must be remitted to NCI CTCAE (Version 5.0) ≤1 degree (except for alopecia or other toxicities that the investigator deems to pose no risk to the patient's safety).

10) Adequate bone marrow functional reserve:

1. White blood cell count (WBC) ≥3.0×10^9 / L
2. Neutrophil count (ANC) ≥1.5×10^9 / L
3. Platelet count (PLT) ≥70×10^9 / L 11) Liver, kidney and heart function tests are basically normal (based on the normal values in the laboratories of each research center) :

a. Total bilirubin (TBIL) ≤3× upper limit of normal (ULN) b. Alanine aminotransferase and aspartate aminotransferase (ALT/AST) ≤2.5×ULN (≤5 ×ULN for patients with liver metastasis) c. Serum creatinine ≤1.5×ULN or creatinine clearance rate (Ccr) ≥60 ml/min; d.Left ventricular ejection fraction (LVEF) ≥ 55%, e. QTcF(Fridericia correction) ≤ 470 ms. 12) Be able to understand the research process, voluntarily participate in this research, and sign the informed consent form.

Exclusion Criteria

If a subject experiences any of the following situations, they will not be eligible to participate in this study:

1. Patients with HR+/ HER2-MBC who have not received endocrine therapy before;
2. Has not received any treatment for metastatic breast cancer;
3. Received more than two chemotherapy regimens for metastatic breast cancer;
4. Patients who are known to be allergic to the active ingredient or other ingredients of the investigational drug.
5. Pregnant or lactating women, and women of childbearing age who refused to take effective contraceptive measures during the study period.
6. Those with severe heart disease or discomfort, expected to be unable to tolerate chemotherapy, including but not limited to: fatal arrhythmia or higher-grade atrioventricular block, unstable angina pectoris, clinically significant valvular heart disease, electrocardiogram showing transmural myocardial infarction, uncontrollable hypertension;
7. Any other circumstances where the researcher deems the patient unsuitable for participation in this study, any concomitant diseases or conditions that may interfere with participation in the study, or any serious medical conditions that may affect the safety of the subjects (such as uncontrollable heart disease, hypertension, active or uncontrollable infection, active hepatitis B virus infection).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival，PFS（Independent Review Committee） | 2 years
  The time from the beginning of treatment to the progression or death of the patient

SECONDARY OUTCOMES:
Progression Free Survival，PFS（Investigator） | 2 years
  The time from the beginning of treatment to the progression or death of the patient
Objective Response Rate，ORR | 2 years
  the proportion of patients with a tumor volume reduction of ≥30% and a minimum timeframe according to accepted response evaluation criteria (e.g., RECIST version 1.1 in solid tumors), including cases of complete response (CR) and partial response (PR).
Clinical Benefit Rate，CBR | 2 years
  Proportion of confirmed complete response, partial response, or stable disease ≥ 24 weeks.
Disease Control Rate， DCR | 2 years
  Proportion of patients with stable or shrinking tumor size，sum of the proportions of complete remission (CR), partial remission (PR) and stable disease (SD)
Overall survival time ，OS | 2 years
  The time from the start of randomization to death due to any cause.
the rate of adverse events | 2 years
  The probability and severity of adverse reactions, and the extent and incidence of AEs were assessed according to CTCAE.
Quality of life scale score，QoL | 2 years
  The function or quality of a patient's physical, psychological, and social adaptability is also known as quality, which is assessed according to the EROTC C30 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jianli Zhao, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat Sen Memorial Hospital，Sun Yat sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
As personal information of patients is involved, we decided not to share individual participant data of patients.

REFERENCES:
- [Background] Litton JK, Rugo HS, Ettl J, Hurvitz SA, Goncalves A, Lee KH, Fehrenbacher L, Yerushalmi R, Mina LA, Martin M, Roche H, Im YH, Quek RGW, Markova D, Tudor IC, Hannah AL, Eiermann W, Blum JL. Talazoparib in Patients with Advanced Breast Cancer and a Germline BRCA Mutation. N Engl J Med. 2018 Aug 23;379(8):753-763. doi: 10.1056/NEJMoa1802905. Epub 2018 Aug 15. PMID 30110579
- [Background] Iglehart JD, Silver DP. Synthetic lethality--a new direction in cancer-drug development. N Engl J Med. 2009 Jul 9;361(2):189-91. doi: 10.1056/NEJMe0903044. Epub 2009 Jun 24. No abstract available. PMID 19553640
- [Background] Robson M, Im SA, Senkus E, Xu B, Domchek SM, Masuda N, Delaloge S, Li W, Tung N, Armstrong A, Wu W, Goessl C, Runswick S, Conte P. Olaparib for Metastatic Breast Cancer in Patients with a Germline BRCA Mutation. N Engl J Med. 2017 Aug 10;377(6):523-533. doi: 10.1056/NEJMoa1706450. Epub 2017 Jun 4. PMID 28578601
- [Background] Gonzalez-Martin A, Pothuri B, Vergote I, DePont Christensen R, Graybill W, Mirza MR, McCormick C, Lorusso D, Hoskins P, Freyer G, Baumann K, Jardon K, Redondo A, Moore RG, Vulsteke C, O'Cearbhaill RE, Lund B, Backes F, Barretina-Ginesta P, Haggerty AF, Rubio-Perez MJ, Shahin MS, Mangili G, Bradley WH, Bruchim I, Sun K, Malinowska IA, Li Y, Gupta D, Monk BJ; PRIMA/ENGOT-OV26/GOG-3012 Investigators. Niraparib in Patients with Newly Diagnosed Advanced Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2391-2402. doi: 10.1056/NEJMoa1910962. Epub 2019 Sep 28. PMID 31562799
- [Background] Ray-Coquard I, Pautier P, Pignata S, Perol D, Gonzalez-Martin A, Berger R, Fujiwara K, Vergote I, Colombo N, Maenpaa J, Selle F, Sehouli J, Lorusso D, Guerra Alia EM, Reinthaller A, Nagao S, Lefeuvre-Plesse C, Canzler U, Scambia G, Lortholary A, Marme F, Combe P, de Gregorio N, Rodrigues M, Buderath P, Dubot C, Burges A, You B, Pujade-Lauraine E, Harter P; PAOLA-1 Investigators. Olaparib plus Bevacizumab as First-Line Maintenance in Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2416-2428. doi: 10.1056/NEJMoa1911361. PMID 31851799
- [Background] Sun C, Yin J, Fang Y, Chen J, Jeong KJ, Chen X, Vellano CP, Ju Z, Zhao W, Zhang D, Lu Y, Meric-Bernstam F, Yap TA, Hattersley M, O'Connor MJ, Chen H, Fawell S, Lin SY, Peng G, Mills GB. BRD4 Inhibition Is Synthetic Lethal with PARP Inhibitors through the Induction of Homologous Recombination Deficiency. Cancer Cell. 2018 Mar 12;33(3):401-416.e8. doi: 10.1016/j.ccell.2018.01.019. PMID 29533782
- [Background] Severson TM, Wolf DM, Yau C, Peeters J, Wehkam D, Schouten PC, Chin SF, Majewski IJ, Michaut M, Bosma A, Pereira B, Bismeijer T, Wessels L, Caldas C, Bernards R, Simon IM, Glas AM, Linn S, van 't Veer L. The BRCA1ness signature is associated significantly with response to PARP inhibitor treatment versus control in the I-SPY 2 randomized neoadjuvant setting. Breast Cancer Res. 2017 Aug 25;19(1):99. doi: 10.1186/s13058-017-0861-2. PMID 28851423
- [Background] Gruber JJ, Afghahi A, Timms K, DeWees A, Gross W, Aushev VN, Wu HT, Balcioglu M, Sethi H, Scott D, Foran J, McMillan A, Ford JM, Telli ML. A phase II study of talazoparib monotherapy in patients with wild-type BRCA1 and BRCA2 with a mutation in other homologous recombination genes. Nat Cancer. 2022 Oct;3(10):1181-1191. doi: 10.1038/s43018-022-00439-1. Epub 2022 Oct 17. PMID 36253484
- [Background] Liu JF, Barry WT, Birrer M, Lee JM, Buckanovich RJ, Fleming GF, Rimel BJ, Buss MK, Nattam SR, Hurteau J, Luo W, Curtis J, Whalen C, Kohn EC, Ivy SP, Matulonis UA. Overall survival and updated progression-free survival outcomes in a randomized phase II study of combination cediranib and olaparib versus olaparib in relapsed platinum-sensitive ovarian cancer. Ann Oncol. 2019 Apr 1;30(4):551-557. doi: 10.1093/annonc/mdz018. PMID 30753272
- [Background] Liu JF, Barry WT, Birrer M, Lee JM, Buckanovich RJ, Fleming GF, Rimel B, Buss MK, Nattam S, Hurteau J, Luo W, Quy P, Whalen C, Obermayer L, Lee H, Winer EP, Kohn EC, Ivy SP, Matulonis UA. Combination cediranib and olaparib versus olaparib alone for women with recurrent platinum-sensitive ovarian cancer: a randomised phase 2 study. Lancet Oncol. 2014 Oct;15(11):1207-14. doi: 10.1016/S1470-2045(14)70391-2. Epub 2014 Sep 10. PMID 25218906